CLINICAL TRIAL: NCT04241120
Title: Feasibility Study for Treating Trichotillomania With Wearable Device and App System Using Habit Reversal Training
Brief Title: Feasibility Study for Treating Trichotillomania With Wearable Device and App System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HabitAware Inc. (Industry)
Collaborators: Marquette University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 31257150; R43MH114773 (NIH)
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-02

CONDITIONS: Trichotillomania
Keywords: Hair Pulling Disorder; Body-Focused Repetitive Behaviors; Trichotillomania
MeSH Terms: conditions — Trichotillomania

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group - HabitAware condition (Experimental): This group will receive the device which alerts the participant when performing hair pulling behavior and the app which provides psychoeducation and components of Habit Reversal Training.
  Interventions: Behavioral: Device and app system designed for participant to self-administer Habit Reversal Training
- Control group - reminder bracelet condition (Placebo Comparator): This group will receive only a device that vibrates randomly several times per hour as a reminder not to pull.
  Interventions: Behavioral: Reminder bracelet control condition

INTERVENTIONS:
Behavioral: Device and app system designed for participant to self-administer Habit Reversal Training — Participants will receive an awareness bracelet and an app that work together to implement key features of Habit Reversal Training. The participant will take part in psychoeducation, awareness training, and competing response training related to trichotillomania.
  Arms: Experimental group - HabitAware condition
Behavioral: Reminder bracelet control condition — Participants will receive a bracelet programmed to vibrate randomly several times per hour during waking hours. They will be instructed this is a reminder not to pull.
  Arms: Control group - reminder bracelet condition

SUMMARY:
Trichotillomania is characterized by recurrent hair pulling resulting in hair loss causing significant distress and impairment which persists despite repeated attempts to stop. Behavioral based therapies focused on increasing awareness of hair pulling followed by the use of an incompatible behavior have proven effective. In an effort to enhance awareness, a wrist worn motion detection device was created. In this study, we will test the feasibility of the HabitAware device and accompanying app as a system for delivering self-administered habit reversal training (HRT).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Speak fluent English
3. Current diagnosis of TTM
4. Score above the normative mean on the automatic pulling subscale of the MIST-A
5. Not on psychotropic medication or on a stable dose (i.e., same dose for past 6 weeks)

Exclusion Criteria:

1. Currently receiving psychotherapy
2. Other psychiatric condition requiring more immediate care
3. Have previously used any behavior awareness devices (e.g. Keen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- HabitAware, Inc., Saint Louis Park, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group - HabitAware Condition | Control Group - Reminder Bracelet Condition
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group - HabitAware Condition | Control Group - Reminder Bracelet Condition | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (15.5) | 31.2 (7.6) | 36.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 5 | 13
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in the HabitAware Condition That Wore the Device for 6 Hours Per Day and More Than 4 Days Per Week.
Description: Measured via post-treatment surveys.
Time Frame: Four weeks
Population: This outcome measure was only for the experimental group.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group - HabitAware Condition | Control Group - Reminder Bracelet Condition
Number analyzed (Participants) | 10 | 0
Participants | 9 | 0

2. Secondary Outcome: Percentage of Participants That Reported the Device >3 on a Scale of 1-5 for Accuracy.
Description: Measured by post treatment survey results
Time Frame: Four weeks
Population: This outcome measure was only for the experimental group.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group - HabitAware Condition | Control Group - Reminder Bracelet Condition
Number analyzed (Participants) | 10 | 0
Participants | 10 | 0

3. Secondary Outcome: Number of Participants That Can Implement HRT Procedures With 80% Accuracy
Description: Measured by trained clinician observing the participant perform the procedures
Time Frame: Four weeks
Population: This outcome measure was only for the experimental group.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group - HabitAware Condition | Control Group - Reminder Bracelet Condition
Number analyzed (Participants) | 5 | 0
Participants | 4 | 0

4. Secondary Outcome: Number of Participants With 30% Improvement in Clinical Symptoms
Description: Measured via pre- and post-treatment MGH-HPS (Massachusetts General Hospital Hair Pulling Scale) and/or NIMH-TSS (National Institute of Mental Health - Trichotillomania Symptom Severity) scores for those in the HabitAware conditions.
Time Frame: Four weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group - HabitAware Condition | Control Group - Reminder Bracelet Condition
Number analyzed (Participants) | 10 | 5
Participants | 6 | 3

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Experimental Group - HabitAware Condition | Control Group - Reminder Bracelet Condition
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT04241120/Prot_SAP_000.pdf